CLINICAL TRIAL: NCT04287231
Title: The Effect of The Five-Session Dual-Transcranial Direct Current Stimulation on Lower-Limb Performance In Sub-Acute Stroke
Brief Title: The Effect of The Five-Session Dual-tDCS On Lower-Limb Performance in Sub-Acute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MU-CIRB 2019/045.1102.1
Record Dates: First submitted 2020-01-09; First posted 2020-02-27 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-tDCS & PT (Experimental): Dual tDCS: the anodal tDCS will be applied over the M1 of the lesioned hemisphere, while the cathodal tDCS will be applied over the M1 of the non-lesioned hemisphere for 20 mins before physical therapy (about 1 hours). Current intensity is fixed at 2 mA and current will flow continuously. Physical therapist will give an intervention program for lower limb performence.
  Interventions: Device: Transcranial direct current stimulation
- Sham-tDCS & PT (Active Comparator): Sham tDCS: the anodal tDCS will be applied over the M1 of the lesioned hemisphere, while the cathodal tDCS will be applied over the M1 of the non-lesioned hemisphere, current intensity will be 2mA (sham mode). Physical therapist will give an intervention program for lower limb performence.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — This instrument will be used to induce post-stroke motor recovery, two different monocephalic montages are typically used to restore excitability in the lesioned hemisphere and to down regulate excitability of the non-lesioned hemisphere and rebalance Interhemispheric inhibition. each participant will undergo a 20-minute period of tDCS, applied at 2 mA through a pair of saline-soaked surface sponge electrodes (35 cm2).

SUMMARY:
The aim of the present study is to determine the effect of the five-session dual-tDCS combine with physical therapy on gait performance, balance and lower limbs muscle strength in patients with subacute stroke.

DETAILED DESCRIPTION:
Stroke is a leading cause of long term disability. The recovery of motor function after stroke is often incomplete, despite classical rehabilitation techniques. In the beginning of the 21st century, transcranial direct current stimulation (tDCS) was introduced as a non-invasive tool to reversibly modulate brain excitability in humans in which a device sends constant low direct current (DC) delivered to the area of interest through the electrodes. Transcranial direct current stimulation (tDCS) has been used in neurorehabilitation to benefit ischemic stroke patients at different stage of stroke especially during acute, sub-acute and chronic phase with positive and safety reports.

After stroke, the excitability of the lesioned hemisphere is decreased and seen like overactive of the excitability of non-lesioned hemisphere. Abnormally high interhemispheric inhibition (IHI) drive from intact to lesioned hemisphere has been reported. The neural plasticity begins in early stages after stroke. Prevent the imbalance IHI and increase the excitability of the lesioned hemisphere in the early phase would be a beneficial for stroke rehabilitation.

Based on the polarity-specific effects, anodal tDCS increases cortical excitability and cathodal tDCS decreases cortical excitability. Transcranial direct current stimulation (tDCS) can be applied in two distinct montages: monocephalic and bi-hemispheric/dual-tDCS (applying two electrodes over both cerebral hemispheres at the same time). To induce post-stroke motor recovery, two different monocephalic montages are typically used: i) to restore excitability in the lesioned hemisphere: anode over the lesioned hemisphere and the cathode as the reference electrode placed over the contra-orbital area ii) to down regulate excitability of the non-lesioned hemisphere and rebalance IHI: cathode over the non-lesioned hemisphere and the anode as the reference electrode. Dual-tDCS can be also applied, permitting simultaneous coupling of excitatory and inhibitory effects on both cortices. There are few evidences showing that tDCS (monocephalic and bi-hemispheric/dual-tDCS) could improve lower limb performance at immediate and at least 3 months. However, there is still unclear effect on gait performance and muscle strength.

Recently, dual-hemisphere tDCS, in which, excites one hemisphere using anodal stimulation and inhibits the other by cathodal stimulation has been described in healthy volunteers to greater enhance hand motor learning compared to uni-hemispheric tDCS. The corresponding tDCS-induced changes were reported in imaging study to involve interhemispheric interactions.

Dual-tDCS has been more recent used in rehabilitation aiming to reduce the inhibition exerted by the non-lesioned hemisphere on the lesioned hemisphere and restore the normal balance of the IHI. Dual-tDCS combined with training or simultaneous occupational/physical therapy has been reported to improve motor skill learning and functions of the paretic upper limb in chronic stroke patients.

Lower-limb functions are commonly disabling after stoke, however, less studies have focused the effect of tDCS on lower limb functions. A single session of anodal tDCS over the lower limb M1 has reported to acutely enhance the effect of motor practice of the paretic ankle, force production of the paretic knee extensors, and postural stability in chronic stroke patients. A study showed an improvement of walking speed immediately after a single session of dual-tDCS alone in sub-acute stroke patients .

Based on the previous study, 1-2 mA current intensity of tDCS is usually used for modulating brain activity. The proper current density delivered is between 0.029-0.008 mA/cm 2. The higher current density, the longer lasting, stronger, and deeper cortical neuron stimulation. Therefore, 2 mA current intensity of tDCS was applied in stroke patients for lower limb performance improvement. Following homologous brain regions, the motor area of lower extremities is in depth and previous studies demonstrated that current intensity 2 mA of tDCS could pass through the lower extremities area of the brain.

Moreover, Tahtis et al, 2013 found that using 2 mA of dual-tDCS could improve walking speed immediately after a single session in sub-acute stroke and Klomjai et al, 2018 found that a single session of dual-tDCS 2 mA with physical therapy in sub-acute stroke immediately improved sit to stand performance greater than physical therapy alone. The mechanisms of actions was hypothesized that when stimulation continuously has effect on neuronal plasticity changes. Therefore, they suggested that further study shall implement more sessions of dual-tDCS combined with physical therapy to improve lower limb performance and determine the long lasting-after effect.

The effect of 5-consecutive sessions dual-tDCS during physical therapy on upper limb performance showed significant improvement of upper limb motor functions and maintained at least 1 week. In this study, long-lasting effect was demonstrated at least one week to three months. There are evidences that 5 consecutive days of uni-hemisphere tDCS appeared to improve lower limb motor functions without serious adverse effects in patients with stroke.It is still unclear for the effect of multiple sessions of dual-tDCS on gait performance and muscle strength as well as the long lasting after-effect of multiple sessions of dual-tDCS.

Therefore, the aim of the present study is to investigate the efficacy of 5 consecutive sessions of dual-tDCS combined with conventional physical therapy on the lower limb functions after stroke in sub-acute. Clinical outcomes for lower limb performance evaluations will consist of muscle strength assessed by hand-held dynamometer, the Time up and go test for lower limb functional performance, Five times sit to stand test for dynamic balance and muscle strength, and the Zebris Force distribution measurement (FDM) for gait analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age range 20-75 years
* First ever-ischemic lesion in the territory of middle cerebral artery or anterior cerebral artery. Diagnostic confirmation will be performed by CT scan or MRI
* Sub-acute onset (1-6 months after the stroke onset)
* Able to walk without physical assistance at least 6 meters

Exclusion Criteria:

* All subjects will be excluded from the study if they have:

  * Not cooperative or cannot understand the instruction
  * Clinical unstable such as vital sign unstable (systolic blood pressure (SBP) ≥ 185 mmHg or diastolic blood pressure (DBP) ≥ 110 mmHg (98) and resting heart rate averaging ≥ 100 bpm (99))
  * No clear neurological antecedent history or psychiatric disorder
  * Moderate pain in any joint of both lower limb (Pain Scale (VAS) ≥ 4/10)
  * Unstable medical conditions such as being in the middle of changing medical treatment.
  * Condition that may increase the risk of stimulation such as epilepsy, pregnancy, unexplained headaches, intracranial metal, pacemaker (evaluating by subjective examination).
  * Participate in the other protocol or receive alternative treatment such as transcranial magnetic stimulation within 1 month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) | 15 minutes
  Force distribution measurement (FDM) will be used to analyze gait cycle. The platform will be detecting the force and weight bearing when foot's patients contact the platform and calculate gait parameter.
  This system was used to analyze gait cycle (step length in cm, step time in second, speed in km/h and cadence in step/minute).
  Participants walked 3 meter per trial on platform and assessed 5 times. The result was selected from average five trials. Participants can rest between trials about 2 minutes or as long as they desired to avoid fatigue.
Timed-up and go test (TUG) | 5 minutes
  The Timed-up & Go (TUG) test is a simple and quick functional mobility test that requires a subject to stand up, walk 3 m, turn, walk back, and sit down.
  The objective of TUG is to determine fall risk and measure the progress of balance, sit to stand, and walking.
  This test was initially designed for elderly persons, but is used for people with Parkinson, stroke, Alzheimer, CVA, Huntington disease and others
  The TUG were assessed only 1 trial and participant were performed as comfortable speed. Materials of TUG are One chair with armrest, stopwatch, tape (to mark 3 meters). The patient starts in a seated position. After that the patient stands up upon therapist's command walks 3 meters, turns around, walks back to the chair and sits down. The time stops when the patient is seated and the subject is allowed to use an assistive device. Be sure to document the assistive device used.
Five Times Sit to Stand Test (FTSTS) | 5 minutes
  The FTSTS measures the functional strength of the lower limbs. Subjects sat with their arms folded across the chest and their back against the chair's backrest. They were asked to stand up fully and sit down again 5 times as quickly as possible. The test was repeated 3 times
  The Five-Times-Sit-to-Stand test (FTSTS) is a clinical test that explores postural control and lower limb muscular strength, devised to accommodate patients who can perform the sit-to-stand activity at least five times. As such, it is a test helpful in quantifying a daily transitional movement while also helping to assess fall risk and disability
  The FTSTS were assessed 2 times and selected score of the best trial. Participants can rest between trials about 2 minutes or as long as they desire to avoid fatigue.

SECONDARY OUTCOMES:
Hand-held dynamometer (HHD) | 15 minutes
  The HHD measures the muscle strength. The HHD is simple, quantitative evaluation and widely used for measurement of muscle strength.
  The strength of lower limbs (hip flexor, hip extensor, hip abductor, knee flexor, knee extensor, ankle dorsiflexor and ankle plantarflexor) were assessed by using the hand-held dynamometer.
  The strength of lower limbs included hip flexor, hip extensor, hip abductor, knee flexor, knee extensor, ankle dorsiflexor and ankle plantarflexor were assessed by using the hand-held dynamometer. Hip flexor,ankle dorsiflexor and ankle plantarflexor was assessed in supine position, knee extensor was assessed in sitting position, hip extensor and knee flexor were assessed in prone position and hip abductor was assessed in side lying position. Each muscle was assessed 2 times and selected score of the best trial. Participants can rest between trials about 1 minute or as long as they desired to avoid fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Wanalee Klomjai, PhD, Study Director — MU
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Nakonpathom, Thailand

IPD SHARING:
Plan to Share IPD: No